CLINICAL TRIAL: NCT01402726
Title: Renal Sympathetic Modification in Patients With Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Jiangsu Provincial People's Hospital (Other); Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuehui Yin, Director and Professor, Dept. of Cardiology, the second affiliated hospital of Chongqing Medical University, Chongqing Cardiac arrhythmias service center, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWAN-HF
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure
Keywords: renal artery; sympathetic nerves; modification; heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- renal sympathetic modification (Experimental): Renal artery ablation to modify sympathetic activity in patients with heart failure.
  Interventions: Procedure: renal sympathetic modification
- Absolute medicine therapy (No Intervention): Maintenance of anti-heart failure medications only

INTERVENTIONS:
Procedure: renal sympathetic modification — Device: THERMOCOOL® Catheter Renal sympathetic modification with a catheter-based procedure
  Other Names: renal denervation
  Arms: renal sympathetic modification

SUMMARY:
The purpose of this study is to observe the incident of composite cardiovascular events after renal sympathetic modification using THERMOCOOL® catheter in patients with heart failure, and evaluate safety and efficacy of the intervention.

DETAILED DESCRIPTION:
Heart failure is a clinical syndrome of chronic cardiac dysfunction, with high morbidity and mortality. Traditional pharmacological therapies are used in clinical practice without breakthrough for long time. Previous studies confirmed that partly blocking sympathetic nerves activity contributed to improve cardiac function in patients with heart failure. Renal ablation with sympathetic modification is a new method which is proved to be effective in decreasing sympathetic nerves activity. The investigators hypothesis that renal sympathetic nerves modification is effective and safe in improving cardiac function. This trial is going to recruit 200 patients (Ablation group VS Control group = 1:1) with a follow-up duration of 3 years. Patients in ablation group will receive additional necessary anti-heart failure drugs besides expectant intervention, and patients in control group will receive appropriate anti-heart failure drugs only. The investigators aim to observe the incident of composite cardiovascular events after renal sympathetic modification using THERMOCOOL® catheter in patients with heart failure, and evaluate safety and efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old, and ≤ 75 years old of age
* more than half a year history of heart failure, except for valvular heart disease
* heart failure patients NYHA Class II III IV
* left ventricular ejection function ≤ 40% or ≥ 45% (that is heart failure with preserved ejection fraction) with Simpson's method
* estimated glomerular filtration rate (eGFR) of ≥ 45mL/min
* is competent and willing to provide written, informed consent to participate in this clinical study

Exclusion Criteria:

* patients with acute heart failure
* patients with acute coronary syndrome
* estimated glomerular filtration rate (eGFR) of < 45mL/min
* has the history of renal restenosis or renal stents implantation
* has experienced AMI (old myocardial infarction is not excluded), unstable angina pectoris, cerebrovascular accidents, and alimentary tract hemorrhage within 3 months
* patients with sick sinus syndrome
* pregnant women
* mental disorders
* patients that have allergy to contrast agent
* patients that do not go with follow-up
* others such as researcher considers it is not appropriate to be included into the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-07 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
composite cardiovascular events | three years
  Comprising myocardial infarction, heart failure, sudden death, cardiogenic death

CONTACTS AND LOCATIONS:
Locations (1):
- 2ndChongqingMU, Chongqing, Chongqing Municipality, China